CLINICAL TRIAL: NCT04421521
Title: Acupuncture for Fibromyalgia Syndrome: An Observational Parallel Groups Study
Brief Title: Acunpuncture for Fibromyalgia Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2717
Record Dates: First submitted 2020-04-28; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-04

CONDITIONS: Acupuncture; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Experimental)
  Interventions: Procedure: Acupuncture
- Standard Therapy Group (No Intervention)

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture with disposable needles will be implemented
  Arms: Acupuncture Group

SUMMARY:
patients suffering from fibromyalgia syndrome according to the criteria of the American College of Rheumatology 2010 will be enrolled. All fibromyalgic patients will be subjected to a further ambulatory visit and if an energy deficiency in the Liver and Spleen Meridians will be identified, according to the Traditional Chinese Medicine rules, acupuncture will be planned. If not, a standard therapy with analgesic drugs will be started. Acupuncture treatment will consist of six weekly sessions. Tricyclic antidepressants, anti-epileptic drugs, selective serotonin reuptake inhibitors and opioids will be used as standard strategy. Pain Scores and Fatigue Impact Scale will be assessed before any treatment and after a 28 days follow-up.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of Fibromyalgia

Exclusion Criteria:

coagulation disorders pregnancy pacemaker Implantable Cardioverter Defibrillator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 28 days after the completion of the treatment
  Numeric Rating Scale from 0 (absence of pain )to 10 (worst pain )